CLINICAL TRIAL: NCT02315274
Title: Pilot Study of Between Visit Interaction to Improve Glycemic Control in Pregnancy With Pre-existing Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yogish C. Kudva, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-003219
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Type 1 Diabetes, Pregnancy
Keywords: Type 1 diabetes; Pregnancy; Glycemic variability; Between visit contact
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Patients were provided help with insulin pump and CGM between visits throughout the pregnancy.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm, remote contact. (Experimental): Between visit remote contact.
  Interventions: Other: Frequent remote contact between clinic visits.

INTERVENTIONS:
Other: Frequent remote contact between clinic visits. — Subjects will upload diabetes device data onto websites. Website data will be reviewed by study team who will provide feedback to patients without clinic visits.

SUMMARY:
Hypothesis:

Increased contact with the diabetes care team throughout pregnancy will lead to improved glucose control during pregnancy.

DETAILED DESCRIPTION:
Patient will have weekly contact through the Mayo Patient On-line Services to send in their blood glucose readings and to receive recommendations back regarding insulin dose changes. Information will be analyzed regarding the magnitude of change in insulin dosing and in glycemic variability.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women with type 1 diabetes utilizing either an insulin pump or multiple daily injection insulin program to manage their diabetes

Inclusion Criteria:

* Female with type 1 diabetes and pregnancy
* EDD prior to November 15, 2014
* 18 years of age and older
* On insulin pump or multiple daily injection insulin program
* Signed patient consent form

Exclusion Criteria:

* Exclusion Criteria:

  * Female with type 1 diabetes and pregnancy under age 18 or older than age 45
  * Female with type 2 diabetes or gestational diabetes and pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Glucose variability | Baseline to 9 months
  Glucose variability represented by multiple measures including mean plasma glucose with standard deviation, high blood glucose index, low blood glucose index and average daily risk range.

SECONDARY OUTCOMES:
Changes is severe hypoglycemia | up to 9 months
  Severe hypoglycemic events

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials